CLINICAL TRIAL: NCT05271812
Title: Professional Supporting and Women's Education for Breastfeeding Promotion: Preliminary Study
Acronym: PSWED
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP210925
Record Dates: First submitted 2022-02-28; First posted 2022-03-09 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Breast Feeding
Keywords: Breastfeeding education; Health promotion; Educational technics
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mothers: All women delivered in the recruitment center
- Staff: All staff working in the labor and delivery areas of the recruiting center.

SUMMARY:
Background The long-term benefits of breastfeeding for newborns and mothers are undeniable and scientifically recognized. Current WHO/UNICEF guidelines suggest increasing exclusive breastfeeding to 75.0% by 2030 worldwide. However, there is substantial heterogeneity in breastfeeding practices around the world. Because while breastfeeding promotion is complex, breastfeeding instructions remain without any educational design in general.

Primary Objective:

- Determine the effectiveness of breastfeeding educations among the nursing mothers during first month after childbirth.

Secondary objectives:

* Identify the theoretical and pedagogical engineering framework the breastfeeding educations proposed in antenatal among nursing mothers and professionals.
* Assess the perceived usefulness of nursing mothers regarding to the educational interventions for breastfeeding management and its frequently complications.
* Assess the perceived usefulness of professionals, regarding to the pedagogical engineering of educational interventions offered to nursing mothers.
* Assess women's competency regarding to the educational interventions for breastfeeding management and its frequently complications.
* Evaluate the organization of educational interventions proposed by professionals.

Method & Results:

The results will be obtained by calculating the mean, standard deviation, median and interquartile range. The Chi-square and Yates' uncorrected and corrected tests will be applied for comparison calculation.

Evaluating criteria for feeling of usefulness and breastfeeding competency will be studied using Likert's four level model, 10-Point numerical scales and short answer questions. The relationships between these variables will be studied by using a sequential mixed method combining interpretative, comprehensive, and explanatory approach.

DETAILED DESCRIPTION:
Promoting breastfeeding, a global public health issue The benefits of exclusive breastfeeding are widely recognized by the scientific community for infants and their mothers. Moreover, its promotion has become a global public health target. According to the World Health Organization (WHO), the global average of exclusive breastfeeding (EBF) has increased from 14% in 1985, to 37% in 2015. The WHO report also notes a disparity about EBF prevalence at birth and at six months.

Guidelines and global positioning to promote breastfeeding WHOs' and UNICEFs' Objective proposed in 2030, 75% of newborns should be exclusively breastfed. This represents 10 million children in the world.

Several measures are recommended: professional commitment, training couples to breastfeed, early and close accompaniment of mothers in breastfeeding initiation and its supporting. WHO proposed an accompanying measure through the Baby-Friendly Hospital Initiative (BFHI) label. This label can be revised every five years.

In France, most maternity are not labelled BFHI. Due a lack of means and human resources. According to the last European commission of the Baby-Friendly Hospital Initiative (BFHI) in December 2019, only 46 maternity out of 498 in France, excluding the military health service, are labeled.

Also, WHO has emphasized communication with Couples, health care breastfeeding skills.

French breastfeeding prevalence evolution in relation to its decisive criteria Since 1995, various surveys in France have shown a clear increase of EBF prevalence at birth. However, the last perinatal survey conducted in 2016 showed a decrease between 2010 and 2016, from 60.3% to 52.2%, with an average EBF of 15 weeks. These progressions are insufficient compared to other northern European countries where exclusive breastfeeding rates at maternity discharge exceed 90%.

Breastfeeding is an individual decision, but many reports incriminate the impact of socio-economic, cultural, and psychological criteria and their interactions in an ecosystemic framework in women decision.

Indeed, the "Epifane study" found a correlation between breastfeeding cessation, age, and lower level of maternal education. The EBF rate among the young mothers with a low socioeconomic level drops from 54% to 35% as early as the first month after the birth. The Elfe survey confirmed that the EBF prevalence is higher in older, managerial mothers with a higher level of maternal education.

Geographical origin is one of the criteria that influence breastfeeding rate at long term. Indeed, mothers from sub-Saharan Africa, North Africa, Asia, and America breastfeed more longer.

For mothers in low socioeconomic status, EBF successful is associated with nurturing mother model, previous experiences, and self-esteem, while for mothers in high socioeconomic status, EBF successful is associated with medical discourses, her own breastfeeding knowledges, and self-training.

The domestic tasks between men and women, women investment in her professional careers, and societal standard are another decisive criterion which produce a heterogeneity of the breastfeeding practices between mothers.

However, the medical supervision of pregnancy and labor, and status of newborn at birth influence the breastfed choice. Regarding to Callahan S, a psychologist, sometimes "over-medicalized" supervision of pregnancies can create a couple dependence state on caregivers for making decision to breastfeed. This dependence creates a cognitive conflict that modifies women behaviors and attitudes concerning her birth and breastfeeding objective.

French recommendations and institutional support for breastfeeding According to the National Nutrition and Health Programs and the French health public recommendations, the breastfeed promoting remains principal measure to prevent childhood inequalities in health. This recommendation gives importance to the mothers and couple education. The objective is to transmit to women "a knowledge to act" with the of breastfeeding knowledge acquisition, the development of breastfeeding skills, self-confidence, and motivation. These new instructions are based on "health literacy", a well-developed concept in the field of public health.

WHO has defined this concept as "the personal characteristics and social resources needed by individuals and communities to access, understand, evaluate and use information and services to make health decisions. In Europe, 12% of people surveyed have inadequate health literacy and 35% have limited health literacy according to the Health Literacy Europe (HLS-EU) results. The level of literacy skills of the French is among the lowest in European countries.

Balanced newborns diet and infants through an EBF and its promotion are the major guidelines of National Nutrition and Health Programs in 2018-2022 and in 2019-2023. Thiers objectives provide for a reinforcement of women accompaniment by perinatal professionals before, during and after pregnancy and during breastfeeding.

However, these objectives do not propose the educational actions or programs to promoting breastfeeding. These organisms do not propose guidelines or means for professionals to achieve these objectives.

BREASTFEEDING PRACTICE AND ITS SUPPORTING Currently, one of the sessions of the Preparation to Birth and Parenthood (PNP) is dedicated to the practice of breastfeeding. Couples can benefit, individually or in groups, in the maternity hospital or at home, from a session dedicated to the practice of breastfeeding.

In the hospital sector, the mapping of the promotion of breastfeeding shows that despite an increase in the number of staff trained to accompany breastfeeding mothers, more than 84% of couples are referred to breastfeeding support networks outside the maternity (PMI, private midwives, associations, networks). Only 32% of Staff declare that they have systematically provided written and oral information to couples on breastfeeding.

After discharge, women can benefit fallow-up. This consists of two or three postnatal visits carried out by midwives. It is about making a health supervision, a mother psychological state and her educational needs. Currently, more than 220,000 women benefit from them, with a majority of primiparous women (60%), multiparous women with two children (25%) and multiparous women with three children (13%). The impact of this program on the promotion of breastfeeding, both in terms of support and in economic impact, has not been studied.

For Women, breastfeed is not a natural practice, and she must be always valued and reassured in her breastfeeding. The importance of the psychoeducational approach about breastfeeding are recognized by the professionals. However, breastfeeding education remains empirical, with a lacks pedagogical engineering. In addition, government recommendation's do not provide benchmarks for this activity, nor do they propose pedagogical means to achieve these objectives.

Focus on educational interventions at the international level An international scoping review was carried out to map the educational interventions used, to identify their pedagogical characteristics, and to promote the choice, implementation, and breastfeeding duration.

This literature review revealed that many interventions begin in the third trimester of pregnancy and end in the postnatal period. The teaching strategies are diverse and combined. An increase breastfeeding duration was noted where the pedagogical objectives aim focused on developing women's knowledge of lactation and its complications and the correct breastfeeding positions. The women breastfeed more longer when education methods based on "socioconstructivist" and cognitivist approaches. Interactive tools have effectively raised women's awareness of breastfeeding value and its continuation at mid-term. the desire to breastfeed and its continuation were found when the learning environment and other criteria such as self-esteem, self-efficacy, and personal motivation were considered by the trainers. Finally, the quality of the caregivers and their competencies were the essential factors for breastfeeding continuation at short and mid-term.

This review also allowed us to observe that professionals rarely refer to pedagogical engineering to guarantee the effectiveness of their educational methods.

DESCRIPTION OF THE ELEMENT(S) OF THE RESEARCH This research is interested in the pedagogical dimension and more specifically on pedagogical engineering existing in the educational interventions and its effect on breastfeeding duration at short term.

This research focuses on three elements:

To identified women and professionals' judgments regarding to the educational interventions. The pedagogical evaluations planned allow to map the education practices and to highlight their pedagogical characteristics through didactic analysis. This is a needs determination in pedagogical engineering.

Measuring women and professional's perception of usefulness and their satisfaction levels could provide additional information to evaluate the perceived usefulness of the educational interventions.

Finally, women competencies and its components, self-efficacy level and self-esteem level are the additional criteria to evaluate breastfeeding education impact among the nursing mother.

ELIGIBILITY:
Inclusion Criteria:

- For nursing mothers: Healthy mothers and healthy new-born Upper 18 years old French speaking Agree to be interviewed in two steps: at day 3 &1 month after the birth.

-For Staff: Agree to be interviewed during study

Exclusion Criteria:

- For nursing mothers: Bottle feeding or mixed breastfeeding. Premature new-born or hospitalised in neonatology ward. Refusing to participate

- For Staff: Refusing to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women who delivered in the Armand Trousseau Maternity
  Staff who working in the Armand Trousseau Maternity
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of breastfeeding educations among mothers during first month after childbirth. | First month after birth
  The proportion of nursing mothers receiving the breastfeeding education.

CONTACTS AND LOCATIONS:
Overall Officials: Mehrnoosh Yazdanbakhsh, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital TROUSSEAU, Paris, Ap-hp, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yazdanbakhsh M, De Andrade V, Spiesser-Robelet L, Gagnayre R. The need for educational intervention for breastfeeding women and the professional practice of midwives in France to promote breastfeeding: A joint explanatory study. Eur J Midwifery. 2024 Dec 11;8. doi: 10.18332/ejm/191176. eCollection 2024. PMID 39664091